CLINICAL TRIAL: NCT00001410
Title: A Phase I and II Study of PEG-Glucocerebrosidase in Patients With Type 1 or Type 3 Gaucher Disease
Brief Title: PEG-Glucocerebrosidase for the Treatment of Gaucher Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940014; 94-M-0014
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-12

CONDITIONS: Gaucher's Disease
Keywords: Recombinant Production; Inherited Disease; Lysosomal Disorder; Inborn Error of Metabolism; Enzyme Replacement Therapy; Glucocerebrosidase; Polyethylene Glycol; Gaucher Disease; Recombinant Enzyme
MeSH Terms: conditions — Gaucher Disease; Genetic Diseases, Inborn; Metabolism, Inborn Errors

INTERVENTIONS:
Drug: Lysodase

SUMMARY:
Gaucher disease is a lysosomal storage disease resulting from glucocerebroside accumulation in macrophages due to a genetic deficiency of the enzyme glucocerebrosidase. It may occur in patients of all ages. The condition is marked by enlargement of the liver and spleen (hepatosplenomegaly), low blood and platelet counts, and bone abnormalities. The condition is passed from generation to generation on via autosomal recessive inheritance. There are actually three types of Gaucher disease.

Type I is the most common form. It is a chronic non-neuronopathic form, meaning the disease does not affect the nervous system. The symptoms of type I can appear at any age.

Type 2 Gaucher disease presents prenatally or in infancy and usually results in death for the patient. Type 2 is an acute neuronopathic form and can affect the brain stem. It is the most severe form of the disease.

Type 3 Gaucher disease is also neuronopathic, however it is subacute in nature. This means the course of the illness lies somewhere between long-term (chronic) and short-term (acute).

Currently there is not a cure for Gaucher disease. Treatment for the disease has traditionally been supportive. In some severely affected patients, bone-marrow transplants have corrected the enzyme deficiency, but it is considered a high-risk procedure and recovery can be very slow. Enzyme replacement therapy is another therapy option and has been approved by the Food and Drug Administration (FDA) for use in type 1 patients.

PEG-glucocerbrosidase is a drug designed to clear out the accumulation of lipid (glucocerebroside) from the blood stream. The drug is actually an enzyme attached to large molecules called polyethylene glycol (PEG). The large molecules of PEG allow the enzyme to remain in the blood stream for long periods of time. By modifying glucocerebrosidase with PEG, it is believed that smaller doses will be required, meaning a reduction in cost for the patient and more convenient administration of the drug. The purpose of this study is to evaluate the effects and safety of enzyme replacement therapy using PEG- glucocerebrosidase for the treatment of Gaucher disease.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the biochemical and therapeutic effects and safety of enzyme replacement therapy using polyethyleneglycol (PEG) modified glucocerebrosidase for the treatment of Gaucher disease and to evaluate the benefit to risk ratio. The study is designed to determine the safety and efficacy in Gaucher patients of recombinantly produced human glucocerebrosidase, which is PEG modified. Parameters to be monitored include hemoglobin, platelet counts, organ size, and extent of bony involvement. Pharmacokinetic, pharmacodynamic, and antibody studies will also be evaluated.

ELIGIBILITY:
Patients must be at least 3 years of age.

Must have a biochemically confirmed (enzyme) and/or genetically confirmed diagnosis of type 1 or type 3 Gaucher disease.

Clinical or laboratory signs suggesting need for therapy which will include at least 2 of the following: hemoglobin less than 11 gm/dl; platelets less than 90,000/mm(3); hepatomegaly and/or splenomegaly.

Patient/Guardian must provide written informed consent.

No pregnant or breast feeding women.

No women/men of reproductive potential unless they agree to use an effective contraceptive method.

No patients treated with alglucerase or imiglucerase during the 6 months prior to study entry.

No patients with the diagnosis of type 2 Gaucher disease.

No patients who have a life-threatening disease or are gravely ill.

No patients who have rapidly progressing fatal illness or concomitant malignancy.

No patients who have a chronic infectious disease including HIV or hepatitis B.

No patients chronically on other medications which may interfere with the drug's metabolism or activity.

No patients who received blood transfusion within a month prior to study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Start 1993-10; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Martin BM, Sidransky E, Ginns EI. Gaucher's disease: advances and challenges. Adv Pediatr. 1989;36:277-306. No abstract available. PMID 2675571
- [Background] Martin BM, Tsuji S, LaMarca ME, Maysak K, Eliason W, Ginns EI. Glycosylation and processing of high levels of active human glucocerebrosidase in invertebrate cells using a baculovirus expression vector. DNA. 1988 Mar;7(2):99-106. doi: 10.1089/dna.1988.7.99. PMID 3282855
- [Background] Rappeport JM, Ginns EI. Bone-marrow transplantation in severe Gaucher's disease. N Engl J Med. 1984 Jul 12;311(2):84-8. doi: 10.1056/NEJM198407123110203. PMID 6377066